CLINICAL TRIAL: NCT05181865
Title: A Phase 1/2a, First-In-Human, Open Label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of FL-301 in Patients With Advanced Solid Tumors
Brief Title: Phase 1/2a Study to Evaluate FL-301 in Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Flame Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FL-301-1001
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Pancreas Cancer; Gastric Cancer; Solid Tumor
Keywords: FL-301; Pancreatic Cancer; Gastric Cancer; GEJ; Gastroesophageal Cancer; Solid Tumor; Claudin 18.2
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1 - Cohort 1 (Experimental)
  Interventions: Drug: 1 mg/kg IV FL-301
- Phase 1 - Cohort 2 (Experimental)
  Interventions: Drug: 3 mg/kg IV FL-301
- Phase 1 - Cohort 3 (Experimental)
  Interventions: Drug: 10 mg/kg IV FL-301
- Phase 1 - Cohort 4 (Experimental)
  Interventions: Drug: 20 mg/kg IV FL-301
- Phase 1 - Cohort 5 (Experimental)
  Interventions: Drug: 30 mg/kg IV FL-301
- Phase 2a - Group 1 (Experimental)
  Interventions: Drug: RP2D, IV FL-301
- Phase 2a - Group 2 (Experimental)
  Interventions: Drug: RP2D, IV FL-301
- Phase 2a - Group 3 (Experimental)
  Interventions: Drug: RP2D, IV FL-301

INTERVENTIONS:
Drug: 1 mg/kg IV FL-301 — N = 1
  Other Names: FL-301
  Arms: Phase 1 - Cohort 1
Drug: 3 mg/kg IV FL-301 — N = 3-6
  Other Names: FL-301
  Arms: Phase 1 - Cohort 2
Drug: 10 mg/kg IV FL-301 — N = 3-6
  Other Names: FL-301
  Arms: Phase 1 - Cohort 3
Drug: 20 mg/kg IV FL-301 — N = 3-6
  Other Names: FL-301
  Arms: Phase 1 - Cohort 4
Drug: 30 mg/kg IV FL-301 — N = 3-6
  Other Names: FL-301
  Arms: Phase 1 - Cohort 5
Drug: RP2D, IV FL-301 — Pancreatic Cancer N = 30
  Other Names: FL-301
  Arms: Phase 2a - Group 1
Drug: RP2D, IV FL-301 — Gastric Cancer (Including GEJ) N = 30
  Other Names: FL-301
  Arms: Phase 2a - Group 2
Drug: RP2D, IV FL-301 — Other Solid Tumors N = 30
  Other Names: FL-301
  Arms: Phase 2a - Group 3

SUMMARY:
This is a Phase 1/2a, first-in-human, open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of FL-301 in patients with advanced cancer.

DETAILED DESCRIPTION:
This is a Phase 1/2a, first-in-human, open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of FL-301 in patients with advanced cancer. The study will consist of 2 phases, Phase 1 and Phase 2a.

In Phase 1, dose escalation will proceed according to a rule-based design methodology. Phase 1 will explore dosing in which a single dose of FL-301 is administered by intravenous (IV) infusion every 2 weeks (Q2W) in 4-week cycles. Patients with measurable advanced solid tumors expressing claudin 18.2 may be enrolled, with the cutoff levels further defined in the eligibility criteria. Dose escalation methodology (modified 3+3 design) will utilize prespecified dose increments.

Once the RP2D has been established, Phase 2a will commence to explore preliminary evidence of antitumor efficacy and confirm the safety of FL-301. The dosing schedule will be explored in up to 3 separate patient groups of approximately 30 patients per group.

Group 1 will include patients with pancreatic cancer; Group 2 will include patients with gastric cancer (including gastroesophageal junction [GEJ]); and Group 3 will include patients with any other solid tumor (primarily non-small cell lung cancer [NSCLC], ovarian, and cholangiocarcinoma with claudin 18.2 expression).

Response and progression will be evaluated in this study using computerized tomography (CT) or magnetic resonance imaging (MRI) imaging per RECIST v1.1. Long-term follow-up (survival and disease status, as applicable) will be conducted up to 18 months or until death, start of new anticancer therapy, end of study, or withdrawal of consent, whichever occurs first.

ELIGIBILITY:
General Inclusion Criteria

Applicable to all patients in both the Phase 1 and Phase 2a parts of the study:

* Histological or cytologically confirmed locally advanced or metastatic solid tumor
* Life expectancy >12 weeks.
* Age ≥18 years.
* ECOG performance status 0 or 1 at screening.
* Fully vaccinated against COVID-19 at least 3 weeks before C1D1. If under consideration for a booster, the booster administration needs to be complete within the same time constraint (ie, at least 3 weeks before C1D1).
* Adequate organ function, defined as:

  * Hematology: defined as absolute neutrophil count (ANC) ≥1.5×109/L, platelet ≥90×109/L, hemoglobin ≥9.0 g/dL (in the absence of transfusion and use of growth factors within the last 14 days of screening labs).
  * Renal function defined as calculated creatinine clearance (CCr) or radioisotope glomerular filtration rate >60 mL/min/1.73 m2 calculated by Cockcroft-Gault formula or normal serum creatinine with a maximum serum creatinine of 1.5 mg/dL.
  * Hepatic Function:

    * Alanine aminotransferase (ALT) ≤2.5 × ULN; ≤5 × ULN if with liver metastases.
    * Total bilirubin ≤1.5×ULN.
  * Serum Electrolytes:

    * Serum potassium, calcium, magnesium, and phosphate within normal limits or not worse than CTCAE v5.0 Grade 1 and asymptomatic. If values are low on the initial screening assessment, supplements may be given, if clinically appropriate, and values repeated to confirm within CTCAE v5.0 Grade 1 limits.

Specific criteria for Phase 1:

* Positive claudin 18.2 tumor expression defined as ≥50% of tumor cells demonstrating moderate-to-strong membranous staining (2+/3+) by IHC assay performed on sections of tumor derived from formalin fixed paraffin block.
* Pathological diagnosis (histological) of any solid tumor cancer with positive claudin 18.2 tumor expression as defined above.

Specific criteria for Phase 2a:

* Positive claudin 18.2 tumor expression defined as ≥70% of tumor cells demonstrating moderate-to-strong membranous staining (2+/3+) by IHC assay performed on sections of tumor derived from formalin fixed paraffin block.
* At least 1 measurable target lesion as defined by RECIST 1.1
* Disease progression or relapse following conventional chemotherapy, patient must have documented radiological progression during or after their most recent anticancer therapy:

  * Pancreatic cancer: Patient should have received at least one but no more than two systemic therapies for their metastatic diseases
  * Gastric cancer (including GEJ cancer): Patient should have received at least two but no more than three systemic therapies for their metastatic diseases;
  * Other solid tumor cancers: Patients with other solid tumors who have no standard therapies available

Exclusion Criteria

Patients who meet any of the following criteria will be excluded:

* History of severe infusion reaction with monoclonal antibody treatment.
* Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening.
* Known history of HIV.
* Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Presence of other active cancers, or history of treatment for invasive cancer ≤3 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, noninvasive) are eligible, as are patients with history of nonmelanoma skin cancer.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Active central nervous system (CNS) disease involvement, defined by cerebrospinal fluid (CSF) cytology, magnetic resonance imaging (MRI) or computerized tomography (CT); patients with asymptomatic CNS metastases are eligible if they have been clinically stable for at least 4 weeks prior to the first dose of study drug and do not require interventions such as surgery, radiation or any corticosteroid therapy for management of symptoms related to CNS disease.
* Pregnant or nursing (lactating) women (Appendix B).
* Patients who received claudin 18.2 targeting agents previously.
* Prior radiotherapy:

  * Non-CNS site of radiation must be completed >2 weeks prior to FL-301 infusion
  * CNS directed radiation must be completed >4 weeks prior to FL-301 infusion as long as patients are asymptomatic post radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Phase 1: The incidence of DLTs (during DLT observation period) | Up to 12 months
  Determine the MTD, and/or to select an RP2D, and investigate the safety and tolerability of FL-301 in patients with advanced solid malignancies
Phase 2a (Expansion): ORR (CR + PR) assessed centrally by RECIST v1.1 | Up to 12 months
  Assess the preliminary antitumor efficacy of FL-301, by central RECIST v1.1

SECONDARY OUTCOMES:
Phase 1: Incidence of patients with TEAEs and SAEs | Up to 12 months
  Characterize the safety and tolerability of FL-301
Phase 1: Incidence of patients who develop ADAs and neutralizing ADAs during treatment with FL-301 | Up to 12 months
  Characterize the immunogenicity of FL-301
Phase 1: ORR (CR + PR), DOR, and DCR assessed locally by RECIST v1.1 | Up to 12 months
  Assess the preliminary antitumor efficacy of FL-301
Phase 1: PK parameters - Cmax | Up to 12 months
  Characterize the PK of FL-301
Phase 1: PK parameters - Tmax | Up to 12 months
  Characterize the PK of FL-301
Phase 1: PK parameters - AUC (0-∞) | Up to 12 months
  Characterize the PK of FL-301
Phase 1: PK parameters - AUC (0-τ) | Up to 12 months
  Characterize the PK of FL-301
Phase 1: PK parameters - Half-life (t1/2) | Up to 12 months
  Characterize the PK of FL-301

OTHER OUTCOMES:
Phase 1 (Exploratory): ORR (CR + PR), DOR, and DCR assessed centrally by RECIST v1.1 | Up to 12 months
  Assess the preliminary antitumor efficacy of FL-301
Phase 1 (Exploratory): Explore the predictive potential of biomarkers measured in blood and/or tumor tissue in response to FL-301 | Up to 12 months
  Explore the predictive potential of biomarkers measured in blood and/or tumor tissue in response to FL-301

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Choe-Juliak, MD, Study Director — Flame Biosciences